CLINICAL TRIAL: NCT01918618
Title: Renal Effects of Levosimendan in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan Braun, MD, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA1-044-13
Record Dates: First submitted 2013-07-26; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Treatment of Left Heart Insufficiency in an Operative Setting of Cardiac Surgery
Keywords: levosimendan; renal effects; cardiac surgery; left heart insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Levosimendan: study group
- No Levosimendan: Control group

SUMMARY:
Recent experimental and clinical data suggest a benefit of levosimendan on the kidney function. Therefore, this retrospective, single center, matched-pairs analysis aimed to investigate whether administration of levosimendan was associated with improved renal function in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery (OPS 5-35 bis 5-37) between 2007 and 2011 followed by postoperative observation on an ICU of the anaesthesiology department of the Charité hospital

Exclusion Criteria:

* Patients younger 18
* Preexisting renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery between 2007 and 2011 followed by postoperative observation on an ICU of the anaesthesiology department of the Charité hospital
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change of plasma creatinine (Difference in renal function) | last available value pre-op (baseline), first available value on post-op day 1, 2, 3 and 4
  Only in patients not requiring renal replacement therapy
Change of urine output after surgery (difference in renal function) | post-op day 1, 2, 3, 4
  Only in patients not requiring renal replacement therapy
Cumulative incidence and duration of hemodialysis (Difference in renal function) | last day of hospital stay

SECONDARY OUTCOMES:
Cumulative Length of stay (hospital and ICU) | last day of hospital stay
In-hospital mortality | last day of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - University Medicine Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Yakut N, Yasa H, Bahriye Lafci B, Ortac R, Tulukoglu E, Aksun M, Ozbek C, Gurbuz A. The influence of levosimendan and iloprost on renal ischemia-reperfusion: an experimental study. Interact Cardiovasc Thorac Surg. 2008 Apr;7(2):235-9. doi: 10.1510/icvts.2007.161356. Epub 2007 Dec 3. PMID 18056154
- [Derived] Balzer F, Treskatsch S, Spies C, Sander M, Kastrup M, Grubitzsch H, Wernecke KD, Braun JP. Early administration of levosimendan is associated with improved kidney function after cardiac surgery - a retrospective analysis. J Cardiothorac Surg. 2014 Nov 18;9:167. doi: 10.1186/s13019-014-0167-8. PMID 25399779